CLINICAL TRIAL: NCT06088797
Title: Exploration of the Role of Vision on Spatial Cognition
Acronym: SpatioCog
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0361
Record Dates: First submitted 2023-10-05; First posted 2023-10-18 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Visual Deficiencies
Keywords: spatial cognition; arithmetic; visual deficiency; blind

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- healthy subjects: First time :WISC V 40 minutes Second time :Completion of the 4 experimental tasks 105 minutes
  Interventions: Other: METRIC COMPARISON Tasks : Tactile PVSE test; Other: METRIC COMPARISON Tasks : Classic PVSE test; Other: Mental imagery task; Other: Proprioceptive spatial representation tasks; Other: Tasks assessing number sense based on relative positions or lengths; Other: WISC V Similarity and Span Test; Other: WISC V Arithmetic subtest
- blind: First time :WISC V 40 minutes Second time :Completion of the 4 experimental tasks 105 minutes
  Interventions: Other: METRIC COMPARISON Tasks : Tactile PVSE test; Other: Mental imagery task; Other: Proprioceptive spatial representation tasks; Other: Tasks assessing number sense based on relative positions or lengths; Other: WISC V Similarity and Span Test; Other: WISC V Arithmetic subtest
- low visual acuity: First time :WISC V 40 minutes Second time :Completion of the 4 experimental tasks 105 minutes
  Interventions: Other: METRIC COMPARISON Tasks : Tactile PVSE test; Other: METRIC COMPARISON Tasks : Classic PVSE test; Other: Mental imagery task; Other: Proprioceptive spatial representation tasks; Other: Tasks assessing number sense based on relative positions or lengths; Other: WISC V Similarity and Span Test; Other: WISC V Arithmetic subtest
- reduced visual field: First time :WISC V 40 minutes Second time :Completion of the 4 experimental tasks 105 minutes
  Interventions: Other: METRIC COMPARISON Tasks : Tactile PVSE test; Other: METRIC COMPARISON Tasks : Classic PVSE test; Other: Mental imagery task; Other: Proprioceptive spatial representation tasks; Other: Tasks assessing number sense based on relative positions or lengths; Other: WISC V Similarity and Span Test; Other: WISC V Arithmetic subtest

INTERVENTIONS:
Other: METRIC COMPARISON Tasks : Tactile PVSE test — Tactile PVSE test The tests are presented in 6 independent booklets, each of which tests a distinct skill: comparison of lengths, comparison of sizes, comparison of obliques, perception of environments, comparison of relative positions in relation to a frame and comparison of relative positions with distractors.
  The assessment sheet presented in a table with the expected answers will allow you to note whether the answers are correct (rating 1) or not (rating 0). A total of the correct answers from all the sub-tests will give a total score.
Other: METRIC COMPARISON Tasks : Classic PVSE test — Classic PVSE test Use of the standardized PVSE test printed on thick white paper in 6 separate booklets each containing a subtest (length, size, oblique, middle, relative position and relative position with distractor)
  The assessment sheet presented in a table with the expected answers will allow you to note whether the answers are correct (rating 1) or not (rating 0). A total of the correct answers from all the sub-tests will give a total score.
  Groups: healthy subjects; low visual acuity; reduced visual field
Other: Mental imagery task — This involves answering questions concerning the position or identity of 2 or 3 objects on the basis of the mental representation of a grid by auditory guidance. Each grid must be constructed mentally with the verbal description of the path and the objects encountered.
Other: Proprioceptive spatial representation tasks — 16 configurations of 3 objects with direct or indirect passive exploration of their relative positions.
  Each grid is presented 3 times with the following 3 questions to which the subject answers yes or no by forced choice
  a single measure of the number of correct answers which will be the sum of the correct answers obtained to each of the 3 questions in the direct vs indirect condition
Other: Tasks assessing number sense based on relative positions or lengths — Pointing exercises on a digital line of 50 cm paper tape: the participant points with his finger to a position on the tape, according to the verbal request of the experimenter
  Measures the intermanual gap during requests for evaluation of 5 times the wand, subtracting the length of a wand, then dividing this length by 2.
Other: WISC V Similarity and Span Test — The Wechsler Intelligence Scale for Children - Fifth Edition, Australian Standard (WISC-V) is an individually administered and comprehensive clinical instrument used to assess the general thinking and reasoning skills of children aged six years to 16 years. Test results include a Full-Scale Intelligence Quotient (IQ) score as well as age-equivalent rankings and scores for Verbal Comprehension, Visual Spatial, Fluid Reasoning, Working Memory and Processing Speed composites
Other: WISC V Arithmetic subtest — The WISC-V is an individually administered, comprehensive clinical instrument for assessing the intelligence of children. The primary and secondary subtests are on a scaled score metric with a mean of 10 and a standard deviation (SD) of 3. These subtest scores range from 1 to19, with scores between 8 and 12 typically considered average.

SUMMARY:
Atypical developpement of spatial cognition has been shown in congenital bindness with some consequences on mathematic learning (Cattaneo et al., 2010) as well as on the mental representation of spatial maps (Thinus-Blanc & Gaunet, 1997). This raises the issue of the role of vision in spatial abilities underlying mathematics and locomotion. These difficulties could also be found in case of partial visual deficiency, like very low visual acuity or large peripheral shrinkage of the visual field.

ELIGIBILITY:
Inclusion Criteria:

For all :

* Aged 12 to 25
* Participant not opposed to the research and parents do not oppose participation in the protocol for minors

For healthy volunteers (normal sighted):

- with typical visual development with correction if needed

For participant with Visual Deficiencies:

* with congenital blindness
* or low visual acuity (between 1/10 and 3/10)
* or with visual field peripheral shrinkage (angle <20°).

Exclusion Criteria:

* General knowledge and working memory skills with a standard score of less than 4
* neurological medical history
* Person deprived of liberty by judicial or administrative decision
* Person subject to a legal protection measure (tutorship, curatorship)

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: participant with Visual Deficiencies monitored in the " Centre Technique Régional pour la Déficience Visuelle" or at the " école spécialisée pour déficients visuels "
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
percentage of correct responses | through study completion, an average of 2 year
  The experimental tasks assess allocentric spatial representations in different modalities with correct responses to spatial vs non spatial questions for the Elementary Spatial Perception test and the mental imagery test.

CONTACTS AND LOCATIONS:
Overall Officials: Laure PISELLA, Dr, Principal Investigator — Equipe Trajectoire du CRNL : INSERM U1028, CNRS UMR 5292)
Locations (1):
- Equipe Trajectoire du CRNL : INSERM U1028, CNRS UMR 5292, Lyon, France